CLINICAL TRIAL: NCT06338852
Title: Awareness of Gynaecologists About Role of Physical Therapy in Genital Prolapse
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Sayed Mohamed Nouh, Physiotherapy researcher, Cairo University
Other Study IDs: 4347
Record Dates: First submitted 2024-03-16; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Genital Prolapse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Socio demographic and evaluation questionnaires — Socio demographic and evaluation questionnaires Used to measure the awareness of gynaecologists about role of physical therapy in genital prolapse

SUMMARY:
The aim of this study will be to detect if there is awareness of gynecologists about the role of physical therapy in genital prolapse.

Physical therapy plays an important role in assessment, prevention and treatment of pelvic floor dysfunction and genital prolapse, it helps to stimulate and strength pelvic floor muscle.

Physical therapy treatments for the pelvic floor may include bladder training, pelvic floor muscles training with or without biofeedback, vaginal cones, electro stimulation or other adjuncts to training.

ELIGIBILITY:
Inclusion Criteria:

-

Gynaecologists in private and government hospitals in Egypt

Exclusion Criteria:

* Gynaecologists with less than 5years experience.

Ages: 29 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: They will be selected from outpatient clinic of (Cairo gynaecological Hospitals).
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2023-03-03 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Socio demographic and evaluation questionnaires | Through study completion, an average of 1 year
  This questionnaires used to detect if there is the awareness of gynaecologists about role of physical therapy in genital prolapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and informed consent form
Supporting Information: Study Protocol, ICF